CLINICAL TRIAL: NCT05327985
Title: STOCI: Three-dimensional Analysis of Obliquus Capitis Inferior Muscle Function in the Rotatory Form of Cervical Dystonia by Means of the Cone Beam Mode CT Scanning :Prospective Cohort Study
Brief Title: Three-dimensional Analysis of Obliquus Capitis Inferior Muscle Function in the Rotatory Form of Cervical Dystonia
Acronym: STOCI
Status: Terminated | Type: Observational
Why Stopped: Lack of inclusions
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JBN_2022_1
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cervical dystonia is the most common form of focal dystonia in adults (50-82%). It manifests itself by a abnormal attitude of the head, intermittent or permanent, due to involuntary contraction of the cervical muscles which appears or is accentuated on the occasion of voluntary movement and maintenance posture. The distribution of dystonic muscles is specific to each patient explaining the diversity of patterns encountered. The therapeutic management of DC is essentially local and symptomatic. It is based on the realization of injections of neuro botulinum toxin (BoNT) targeting target (dystonic) muscles responsible for involuntary movements or posture abnormal. Identifying the muscles involved is a step prerequisite for therapeutic intervention.The obliquus capitis inferior (OCI) also known as Lower Oblique belongs to the group of suboccipital muscles.It is the only suboccipital muscle that does not attach to the skull. Its unilateral contraction causes ipsilateral rotation of C1 therefore of the head. The length of the transverse process of the atlas gives it considerable rotary efficiency. It is described as the cephalic rotation starter muscle. It would perform the 30 first degrees of rotation. The rotation of the whole column cervical would then be continued by the synergistic action of the muscle contralateral sternocleidomatoid and Spl. ipsilateral. The level of joint complex C1-C2 the amplitude of rotation corresponds to approximately 50% of the total rotation of the cervical spine. In order to better understand the part played by the OCI muscle in the disorganization of posture and cervical movements in the axial plane (plane of rotation) in the rotary DC, the investigators want biomechanically analyze its function in pathological situation. The physiology of this muscle is richly documented in healthy subjects. But does this knowledge apply in DC? Acquisition of imagery by the "Cone Beam" or CBCT system (Cone Beam Computed Tomography) before and 5 weeks after the injection of BoNT, will allow the analysis of the displacement of each vertebrate.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 70
* Presenting with a diagnosed focal CD with predominantly rotational by a neurologist specialized in abnormal movements
* Receiving botulinum toxin injection at OIC level as part of his treatment
* Express consent to participate in the study
* Member of or beneficiary of a social security scheme

Exclusion Criteria:

* Mobile DC (scrapie and/or myoclonic) that cannot be controlled the recording time by the CBCT system
* Having already benefited from an injection of BoNT as part of their DC in the last three months
* Inability to sit still
* Neurological condition other than DC (parkinsonian syndrome typical or atypical, others.)
* Severe neck pain
* Known or suspected trauma or pathology of the cervical spine, other than DC, having required treatment in the last 6 month
* Same old surgery of the cervical spine
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding women (a urine pregnancy test will be carried out in women under 50)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from predominantly rotatory focal cervical dystonia will be identified directly by investigators at the Fondation A. de Rothschild Hospital during abnormal movement consultations or during specialized rehabilitation sessions.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Changes in posture and main movement rotation of the cervical spine | Before (day0) and after injection of BoNT (after 8 weeks max)
  Movement of primary rotation of the cervical spine on CBCT imaging will be described using the symmetry index (SI), based on the difference angular (in degrees) of the active amplitude of right rotation and left

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre Bleton, Principal Investigator — Hopital Fondation Adolphe de Rothschild
Locations (1):
- Hopital Fondation Adolphe de Rothschild, Paris, France